CLINICAL TRIAL: NCT03317158
Title: PhAse 1/2 StuDy of Modern ImmunotherApy in BCG-Unresponsive, BCG-RelaPsing, and High-Risk BCG-Naive Non-muscle Invasive UroThelial Carcinoma of the BLADDER
Brief Title: Modern Immunotherapy in BCG-Unresponsive, BCG-Relapsing and High Risk BCG-Naive Non-Muscle Invasive Urothelial Carcinoma of the Bladder
Acronym: ADAPT-BLADDER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Noah Hahn, M.D. (Other)
Collaborators: AstraZeneca (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Noah Hahn, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU16-243
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: non-muscle invasive bladder cancer; BCG; immunotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — durvalumab; Gemcitabine; Docetaxel; tremelimumab

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Phase 1: Cohort 1 (Experimental): Durvalumab monotherapy
  Interventions: Drug: Durvalumab (Cohort 1-3)
- Phase 1: Cohort 2 (Experimental): Durvalumab plus BCG
  Interventions: Drug: Durvalumab (Cohort 1-3); Biological: Bacillus Calmette-Guérin (BCG)
- Phase 1: Cohort 3 (Experimental): Durvalumab plus External Beam Radiotherapy (EBRT)
  (BCG re-treatment) - Cross-over to Durvalumab Monotherapy
  Interventions: Drug: Durvalumab (Cohort 1-3); Radiation: External Beam Radiotherapy (EBRT)
- Phase 1: Cohort 4 (Experimental): Durvalumab + Gemcitabine/Intravesical Docetaxel (Gem/Doc)
  The sequence of administration is flexible to allow for scheduling of both the infusion and intravesical treatments.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Durvalumab (Cohort 4/5)
- Phase 1: Cohort 5 (Experimental): NOTE: Cohort 5 was abandoned prior to any patients enrolled.
  Durvalumab + Tremelimumab + Gem/Doc
  The sequence of administration is flexible to allow for scheduling of both the infusion and intravesical treatments. For the intravenous medications, durvalumab should be administered first followed by tremelimumab.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Biological: Tremelimumab; Drug: Durvalumab (Cohort 4/5)
- Phase 1: Cohort 6 (Experimental): Additional Regimens (to be determined)
  Interventions: Other: To be determined
- Phase 2: Cohort 4 Expansion (Experimental): Durvalumab + Gemcitabine/Intravesical Docetaxel (Gem/Doc)
  The sequence of administration is flexible to allow for scheduling of both the infusion and intravesical treatments.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Durvalumab (Cohort 4/5)

INTERVENTIONS:
Drug: Durvalumab (Cohort 1-3) — Durvalumab 1120 mg intravenously Day 1 every 21 days x 8 cycles.
  Other Names: Imfinzi
  Arms: Phase 1: Cohort 1; Phase 1: Cohort 2; Phase 1: Cohort 3
Radiation: External Beam Radiotherapy (EBRT) — EBRT 6 Gy x 3; Cycle 1 Day 1, 3, and 5
  Arms: Phase 1: Cohort 3
Biological: Bacillus Calmette-Guérin (BCG) — Dose level 0 (starting dose) = Full-dose
  Dose level-1 = 1/3rd-dose BCG. Dose level -1 is expected to be utilized during the phase II portion of the study due to the ongoing and persistent shortage of BCG in the US.
  Arms: Phase 1: Cohort 2
Drug: Gemcitabine — Gemcitabine 1000 mg intravesical weekly (+/- 2 days) x 6 doses
  Other Names: Gemzar
  Arms: Phase 1: Cohort 4; Phase 1: Cohort 5; Phase 2: Cohort 4 Expansion
Drug: Docetaxel — Docetaxel 37.5 mg intravesical weekly (+/- 2 days) x 6 doses.
  Other Names: Taxotere
  Arms: Phase 1: Cohort 4; Phase 1: Cohort 5; Phase 2: Cohort 4 Expansion
Biological: Tremelimumab — Tremelimumab 75 mg intravenously Day 1 (+/- 2 days) every 28 days x 4 cycles.
  Arms: Phase 1: Cohort 5
Drug: Durvalumab (Cohort 4/5) — Durvalumab 1500 mg intravenously Day 1 (+/- 2 days) every 28 days x 6 cycles.
  Other Names: Imfinzi
  Arms: Phase 1: Cohort 4; Phase 1: Cohort 5; Phase 2: Cohort 4 Expansion
Other: To be determined — Other regimens to be determined
  Arms: Phase 1: Cohort 6

SUMMARY:
Upon successful screening and registration, enrollment to durvalumab monotherapy (cohort 1) will begin. If DLT criteria outlined in the protocol are exceeded with durvalumab monotherapy (cohort 1), the study will close. Provided the safety of durvalumab monotherapy is established, enrollment to combination regimen cohorts will proceed. Cohorts will simultaneously enroll in parallel to each other with patients assigned to cohorts based on patient slot availability and study site choice of radiation arm participation. Patient assignment to future phase 1 arms would proceed similarly.

Within BCG-containing cohorts, treatment will begin at full-dose BCG. If DLT criteria outlined in Section 5.1.4 are exceeded with full-dose BCG, a one level dose reduction of BCG will be implemented. If DLT criteria outlined in Section 5.1.4 are exceeded with reduced-dose BCG, the BCG-containing cohort will not proceed to Phase 2 of the study. Similarly, if DLT criteria outlined in Section 5.1.4 are exceeded within non-BCG containing cohorts, the non-BCG containing cohort will not proceed to phase 2 of the study. Due to the prolonged half-life of antibody therapies, no dose adjustments are planned for durvalumab in any of the cohorts.

ELIGIBILITY:
Inclusion Criteria (All Patients):

Subject must meet all of the following applicable criteria to participate in this study:

* Histologically confirmed non-muscle invasive urothelial carcinoma of the bladder (Ta, T1, or Tis stage) on TURBT obtained within 60 days of registration.

NOTE: Mixed histologies are permitted, provided a component of urothelial carcinoma is present. Patients with histologically confirmed non- muscle invasive urothelial carcinoma of the bladder (Ta, T1, or Tis stage) on prior TURBT who undergo re-resection of the tumor base to confirm the diagnosis and/or exclude the presence of muscle-invasive disease (T2 or greater) who do not have appreciable tumor in the re-resection TURBT are eligible to enroll provided their re-resection was obtained within 60 days of registration and they meet all other eligibility criteria.

* ECOG (WHO) performance status 0 or 1
* Age ≥ 18 years old at time of consent
* Adequate hematologic, hepatic, and renal function as defined by the following laboratory parameters:

  * White blood cell count (WBC) > 3.0 K/mm3
  * Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
  * Platelets ≥ 100 K/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * ALT and AST ≤ 2.5 x ULN
  * Serum creatinine clearance (CrCl) ≥ 30 mL/min using the modified Cockcroft- Gault equation
* Subjects who give a written informed consent obtained according to local guidelines

Inclusion Criteria (Phase 1 Only):

In addition to the inclusion criteria required of all patients above, the following inclusion criteria are also required of patients enrolling to Phase 1 of the study.

• BCG-unresponsive disease defined by any of the following:

* Persistent or recurrent CIS with or without the presence of concurrent Ta or T1 tumors within 12 months of completion of adequate BCG therapy
* Recurrent high-grade Ta or T1 tumors within 6 months of completion of adequate BCG therapy.

NOTE: In recognition of the fact that procedure scheduling factors beyond the control of the patient or treating physician may cause unintended delays in disease evaluations, patients with pure papillary tumors (Ta or T1) with no components of CIS with recurrence documented within 9 months of completion of adequate BCG therapy who meet all other eligibility criteria may be considered for enrollment after consultation with the study chair.

* Persistent T1 high-grade tumors at the first disease evaluation (e.g. 3- month post-treatment evaluation) following an adequate BCG induction course
* Prostatic urethra involvement of NMIBC
* Adequate BCG therapy is defined as at least one of the following:

  * At least 5 of 6 doses of an initial induction BCG course plus at least 2 of 3 doses of maintenance therapy
  * At least 5 of 6 doses of an initial induction BCG course plus at least 2 of 6 doses of a second induction course.

NOTE: Patients with concurrent non-muscle invasive tumors (CIS, Ta, T1) in the prostatic urethra and/or concurrent non-invasive tumors (CIS, Ta) in the upper urinary tracts (ureter, renal pelvis) are permitted to enroll in Phase 1 of the study. Patients with concurrent T1 tumors in the upper urinary tracts (ureter, renal pelvis) are not eligible to enroll in Phase 1 of the study. Patients who have met the BCG-unresponsive criteria at any time point in their treatment history are permitted to enroll in Phase 1 of the study regardless of the time frame between their most recent BCG treatment administration and study registration dates.

Inclusion Criteria (Phase 2 Only):

In addition to the inclusion criteria required of all patients above, the following inclusion criteria are also required of patients enrolling to Phase 2 of the study.

• High-risk NMIBC defined according to modified EORTC risk criteria summarized as follows:

NOTE: Intermediate- and Low-risk tumors as defined below are not eligible. NOTE: Patients with concurrent non-muscle invasive tumors (CIS, Ta, T1) in the prostatic urethra are permitted to enroll in Phase 2 of the study. At least half of the subjects enrolled to each cohort must have a component of CIS present.

* Low-risk Tumors: Initial or recurrent tumor > 12 months after resection with all of the following:

  --- Solitary tumor

  --- Low-grade
  * < 3 cm
  * No CIS
* Intermediate-Risk Tumors

  --- All tumors not defined in the two adjacent categories (between the category of low and high risk)
* High-risk Tumors. Any of the following:

  * T1 tumor
  * High-grade
  * CIS
  * Multiple and recurrent and large (> 3 cm) Ta low-grade tumors (all conditions must be met for this point on Ta low-grade tumors)

    • BCG-unresponsive, BCG-relapsing, BCG-persistent, or high-risk BCG-naïve NMIBC defined as follows:

NOTE: Patients enrolling to phase 2 will enroll separately into a maximum of three expanded cohorts defined by the BCG exposure population eligibility criteria defined below (BCG-unresponsive, BCG-relapsing, BCG-persistent, and high-risk BCG-naïve). The three possible cohorts for each regimen expanded to phase 2 enrollment will be: BCG-unresponsive, BCG-relapsing and/or BCG-persistent (combined within a single cohort), and high-risk BCG-naïve. It is not anticipated that all three possible phase 2 expansion cohort populations will be pursued for every regimen entering phase 2 expansion. Questions regarding phase 2 expansion cohort populations and patient eligibility should be directed to the study chair. The individual eligibility for phase 2 expanded cohorts according to BCG exposure history are summarized below.

o BCG-unresponsive NMIBC phase 2 expanded cohort. BCG-unresponsive NMIBC is defined by any of the following:

* Persistent or recurrent CIS with or without the presence of concurrent Ta or T1 tumors within 12 months of completion of adequate BCG therapy
* Recurrent high-grade Ta or T1 tumors within 6 months of completion of adequate BCG therapy.

NOTE: In recognition of the fact that procedure scheduling factors beyond the control of the patient or treating physician may cause unintended delays in disease evaluations, patients with pure high-grade papillary tumors (Ta or T1) with no components of CIS with recurrence documented within 9 months of completion of adequate BCG therapy who meet all other eligibility criteria may be considered for enrollment after consultation with the study chair.

* Persistent T1 high-grade tumors at the first disease evaluation (e.g. 3-month post-treatment evaluation) following an adequate BCG induction course
* Prostatic urethra involvement of NMIBC o Adequate BCG therapy is defined as at least one of the following:
* At least 5 of 6 doses of an initial induction BCG course plus at least 2 of 3 doses of maintenance therapy
* At least 5 of 6 doses of an initial induction BCG course plus at least 2 of 6 doses of a second induction course

  * BCG-relapsing and/or BCG-persistent NMIBC phase 2 expanded Cohort. BCG-relapsing and/or BCG-persistent NMIBC is defined by either of the following:

    • BCG-relapsing NMIBC is defined as recurrent high-risk NMIBC after achievement of a complete response to BCG induction therapy which does not meet any of the BCG-unresponsive criteria outlined in the protocol.
  * BCG-persistent NMIBC is defined as persistent high-risk NMIBC at the first disease evaluation after initial BCG induction therapy (with no intervening achievement of complete response) for which a second course of BCG induction therapy is considered a standard of care (e.g. CIS or high grade Ta tumors) which does not meet any of the BCG-unresponsive criteria outlined in the protocol.
  * High-risk BCG-naive NMIBC cohort. High-risk BCG-naive NMIBC is defined as high-risk NMIBC in a patient that has never received intravesical BCG therapy. NOTE: Patients who satisfy the above definition of BCG-unresponsive NMIBC continue to be considered BCG-unresponsive regardless of the receipt of any intervening or additional non-BCG based intravesical therapies (e.g. chemotherapy, non-BCG investigational agents)

Primary Exclusion Criteria:

Exclusion Criteria (All Patients):

* Subjects with muscle-invasive (i.e. T2, T3, T4) locally advanced unresectable, or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within 60 days prior to study registration. The required radiographic imaging includes:

  * Abdomen/Pelvis - CT scan
  * Chest - chest x-ray or CT scan
* Subjects with another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer. Subjects that have completed all necessary therapy and are considered to be at less than 30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment.
* Subjects who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy.
* Any unresolved toxicity NCI CTCAE v4.03 for Cohorts 1-3 and v5.0 for cohorts 4-6 Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by- case basis after consultation with the sponsor-investigator.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the sponsor-investigator.
* Subjects who have received prior therapy with PD-1, PD-L1, or CTLA-4 directed agents.
* Subjects who have had any prior radiation to the prostate or pelvis.

NOTE: The exclusion of patients who have had any prior radiation to the prostate or pelvis applies to both phase 1 and 2 of the trial only within radiation containing study regimens. Patients with a prior history of prostate or pelvic radiation who meet all other eligibility criteria may be considered for phase 1 and phase 2 enrollment to non-radiation containing study regimens after consultation with the study chair.

* Subjects who have undergone major surgery (e.g. intra-thoracic, intra- abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or subjects who have had minor procedures (i.e. TURBT), percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Subjects with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Clinically significant cardiac diseases, including any of the following:

    * History or presence of serious uncontrolled ventricular arrhythmias
    * Clinically significant resting bradycardia
    * Any of the following within 3 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)
    * Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s)
  * Cirrhosis
  * Active Infection (includes chronic active and chronic persistent) --- Tuberculosis --- Hepatitis B (known positive HBV surface antigen (HbsAg). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible

    --- Hepatitis C. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

    --- Known diagnosis of human immunodeficiency virus (HIV/positive HIV 1/2 antibodies) infection (HIV testing is not mandatory)
  * Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    --- Patients with vitiligo or alopecia

    --- Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement

    --- Any chronic skin condition that does not require systemic therapy

    --- Patients without active disease in the last 5 years may be included but only after consultation with the study physician

    --- Patients with celiac disease controlled by diet alone
  * Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
  * Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted. For questions, please consult the sponsor-investigator.
* Pregnant or breast-feeding women. Women of child-bearing potential must have a negative serum test ≤ 14 days prior to starting study drug.
* Women of child-bearing potential, who are biologically able to conceive, and not employing contraception as described in the protocol.
* Fertile males not willing to use contraception, as stated in the protocol.
* Subjects unwilling or unable to comply with the protocol
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

NOTE: Patients, if enrolled, should not receive live vaccine whilst receiving study drugs and up to 30 days after the last dose of study drug.

• Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

3.2.2 Exclusion Criteria (Cohorts 4 and 5 Only)

• Subjects who have received prior intravesical therapy with BOTH gemcitabine and docetaxel

NOTE: Patients who have received either intravesical gemcitabine or intravesical docetaxel (or other taxanes) but not both remain eligible. For example, patients receiving post-TURBT single dose intravesical gemcitabine administration are eligible. Similarly, patients treated with intravesical gemcitabine induction and/or maintenance are eligible. While we typically do not see patients treated with intravesical docetaxel (or other taxanes) monotherapy, if such a patient were identified and screened, they would be eligible. Patients who have received treatment with separate courses of intravesical gemcitabine monotherapy and intravesical docetaxel (or other taxanes) monotherapy are not eligible, unless such therapies occurred more than 24 months ago.

Exclusion Criteria (Phase 1 Only) In Phase 1 of the study, there are no additional exclusion criteria beyond those described of all patients above.

Exclusion Criteria (Phase 2 Only) In addition to the exclusion criteria described of all patients above, the following exclusion criteria apply to patients enrolling to Phase 2 of the study.

• Subjects with concurrent upper urinary tract (i.e. ureter, renal pelvis) high-grade urothelial carcinoma. NOTE: Subjects with concurrent low-grade non-invasive (Ta) upper urinary tract urothelial carcinoma are eligible. Similarly, patients with a history of high-grade upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the recommended phase 2 dose (RP2D) from BCG-unresponsive non-muscle invasive bladder cancer (NMIBC) | 6 months
  Determine the recommended phase 2 dose (RP2D) from BCG-unresponsive non-muscle invasive bladder cancer (NMIBC) patients treated with each of the following immunotherapy study regimens:
  Durvalumab (cohort 1)
  Durvalumab + intravesical BCG (cohort 2)
  Durvalumab + radiation (cohort 3)
  Durvalumab + intravesical Gemcitabine + intravesical Docetaxel (cohort 4)
  Durvalumab + Tremelimumab + intravesical Gemcitabine + intravesical Docetaxel (cohort 5)
  The RP2D of each immunotherapy study arm is defined as the dose level at which < 2 out of 6, < 4 out of 9, or < 5 out of 12 patients enrolled within an individual study arm experience dose-limiting toxicity. Additional details provided in the protocol.
Phase 2: Determine the complete response rate within individual phase 2 expansion cohorts of BCG-unresponsive, BCG-relapsing/persistent, and high-risk BCG-naïve NMIBC subjects treated with each study regimen | 6 months
  The complete response rate within each study arm is defined as the proportion of patients within each arm that demonstrate no evidence of recurrent or persistent high grade urothelial carcinoma of the bladder of any stage at any post-treatment disease assessment.

SECONDARY OUTCOMES:
Phase 1: Assess Adverse Events | 6 months
  The safety profile of BCG-unresponsive NMIBC subjects treated within each study regimen will be assessed by NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 for Cohorts 1-3 and v5.0 for Cohorts 4-6.
Phase 1: Characterize the complete response rate of BCG-unresponsive NMIBC subjects treated with each study regimen | 2 years (24 months)
  The complete response rate within each study arm is defined as the proportion of patients within each arm that demonstrate no evidence of recurrent or persistent high grade urothelial carcinoma of the bladder of any stage at any post-treatment disease assessment.
Phase 1: Characterize the 12-month recurrence free survival (RFS) rate of BCG-unresponsive NMIBC subjects treated with each study regimen | 12 month
  The 12-month RFS rate of BCG-unresponsive NMIBC subjects treated within each study regimen is defined as the proportion of patients within each arm with no evidence of recurrent high grade urothelial carcinoma of the bladder of any stage at the 12-month post-treatment disease assessment.
Phase 2: Determine the 12-month RFS rate within individual phase 2 expansion cohorts of BCG-unresponsive, BCG-relapsing/persistent, and high-risk BCG-naive NMIBC subjects treated with each study regimen | 12 months
  The 12-month RFS rate of BCG-unresponsive, BCG-relapsing/persistent, and high-risk BCG-naive NMIBC subjects treated within each arm is defined as the proportion of patients within each arm with no evidence of recurrent high grade urothelial carcinoma of the bladder of any stage at the 12-month post-treatment assessment.
Phase 2: Identify significant associations between complete response rates and 12-month RFS rates and baseline tumor immunohistochemistry staining patterns of PD-L1 and other relevant mechanism of action targets for each study regimen | 12 months
  Associations between complete response rate and 12-month RFS rates will be assessed by baseline tumor immunohistochemistry staining patterns of PD-L1 (assessed by the SP263 PD-L1 antibody) and other relevant mechanism of action targets for each drug.
Phase 2: Assess Adverse Events | 6 months
  The safety profile within individual phase 2 expansion cohorts of BCG-unresponsive, BCG-relapsing/persistent, and high-risk BCG-naive NMIBC subjects treated within each study arm will be assessed by NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 for Cohorts 1-3 and v5.0 for Cohorts 4-6.

CONTACTS AND LOCATIONS:
Overall Officials: Noah M. Hahn, MD, Principal Investigator — Hoosier Cancer Research Network
Locations (12):
- United States (12):
  - BCG Oncology, Phoenix, Arizona
  - Stanford University, Stanford, California
  - Rush University Medical Cneter, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://hoosiercancer.org